CLINICAL TRIAL: NCT04121351
Title: Physiological Demands Related to Exercises in Singing for Lung Health: A Pilot Study (PHRESH Study)
Brief Title: Physiological Demands Related to Exercises in Singing for Lung Health
Acronym: PHRESH
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic meant continuation of the study was unfeasible at this time.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: ICREC ref:19IC5429
Record Dates: First submitted 2019-09-30; First posted 2019-10-09 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Lung Health; Exercises
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Singing participation — Participants will follow a 15 minute protocol consisting of the components of a Singing for Lung Health class, and a short period walking on a treadmill.

SUMMARY:
This study will assess the physiological demands related to Singing for Lung Health participation.

DETAILED DESCRIPTION:
This study will assess the physiological demands experienced by healthy volunteers participating in components of a Singing for Lung Health session. Oxygen consumption, heart rate, and fixed body sensor output puts related to balance and movement intensity will be assessed. The same parameters will also be assessed during walking on a treadmill at different speeds for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Able to undertake singing components
* Able to undertake walking test
* No contraindications to exercise
* No contraindications to spirometry as per American Thoracic Society/European Respiratory Society criteria
* Capacity to consent to exercise testing.

Exclusion Criteria:

* Any health condition that would preclude them from singing or impede physical activity
* Inability to comply or follow singing exercise instructions
* Active musculoskeletal disease impairing exercise.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption in mL per kilogram per minute during different components of Singing for Lung Health(physical warm up, rhythm exercises, pitch exercises, vocal exercises, repertoire and relaxation) | Single assessment at baseline.
  Assessed using portable metabolic measurement equipment (Oxycon Mobile made by Vyaire).

SECONDARY OUTCOMES:
Heart rate during different components of Singing for Lung Health (physical warm up, rhythm exercises, pitch exercises, vocal exercises, repertoire and relaxation). | Single assessment at baseline.
  Assessed using a portable heart rate monitor.
Comparison of oxygen consumption, in mL per kilogram per minute, achieved during each component of Singing for Lung Health with walking at different speeds | Single assessment at baseline.
  Oxygen consumption, in mL per kilogram per minute, will be assessed during different components of Singing for Lung Health(physical warm up, rhythm exercises, pitch exercises, vocal exercises, repertoire and relaxation. This will be compared with oxygen consumption while walking at three speeds on a treadmill (slow, medium and brisk). Oxygen consumption will be assessed using portable metabolic measurement equipment (Oxycon Mobile made by Vyaire).
Movement intensity during different components of Singing for Lung Health(physical warm up, rhythm exercises, pitch exercises, vocal exercises, repertoire and relaxation). | Single assessment at baseline.
  Assessed with the McRoberts fixed-body sensor MoveTest device.
Changes in centre of mass during different components of Singing for Lung Health (physical warm up, rhythm exercises, pitch exercises, vocal exercises, repertoire and relaxation). | Single assessment at baseline
  Assessed with the McRoberts fixed-body sensor MoveTest device.

CONTACTS AND LOCATIONS:
Overall Officials: Keir Philip, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not currently decided.

REFERENCES:
- [Derived] Philip KE, Lewis A, Buttery SC, McCabe C, Manivannan B, Fancourt D, Orton CM, Polkey MI, Hopkinson NS. Physiological demands of singing for lung health compared with treadmill walking. BMJ Open Respir Res. 2021 May;8(1):e000959. doi: 10.1136/bmjresp-2021-000959. PMID 34045239